CLINICAL TRIAL: NCT06606912
Title: Predictive Effect of Abdominal Fat and Muscle Area Calculated Based on Abdominal CT on Short- and Long-term Outcomes in Patients with Gastric Cancer
Brief Title: Predictive Effect of Abdominal Fat and Muscle Area Calculated Based on Abdominal CT on Gastric Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dong Peng, Dr., First Affiliated Hospital of Chongqing Medical University
Other Study IDs: ZZ2024-158-01
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Gastric Cancers; Colorectal Cancer; Sarcopenia; Obesity and Overweight
Keywords: Subcutaneous Fat; Visceral fat; gastrointestinal cancer; sarcopenia; surgery
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Sarcopenia; Obesity; Overweight; Gastrointestinal Neoplasms | interventions — Adiposity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Skeletal muscle, subcutaneous fat and visceral fat area — CT-based measurement of skeletal muscle, subcutaneous fat and visceral fat areas at L1, L2, L3, L4 and L5 levels.
  Other Names: Sarcopenia; obesity; overweight

SUMMARY:
This study aims to create a clinical prediction model. Abdominal fat and muscle area also play an important role in the prediction of surgical outcomes in colorectal cancer. Studies have shown that excess visceral fat and low skeletal muscle mass (sarcopenia) are associated with poorer postoperative outcomes, including a higher risk of postoperative complications and lower survival. Preoperative imaging techniques such as CT, MRI and ultrasound that provide accurate measurements to assess abdominal fat and muscle area can help surgeons develop individualized surgical and rehabilitation plans, improve surgical success, reduce complications and improve long-term patient prognosis. In this study, the investigators expected to construct a prediction model of abdominal fat and muscle area on the short- and long-term outcomes of gastric and colorectal cancer patients by calculating the abdominal fat and muscle area in different levels of abdominal CT images, in order to further adjust and guide the treatment plan.

DETAILED DESCRIPTION:
This is a retrospective observational study, which is expected to include patients diagnosed with gastric cancer and undergoing radical gastric cancer surgery in the Department of Gastrointestinal Surgery of the First Affiliated Hospital of Chongqing Medical University, the Department of Gastrointestinal Surgery of the Second Affiliated Hospital of Chongqing Medical University, the Department of Gastrointestinal Surgery of the Affiliated Yongchuan Hospital of Chongqing Medical University, and the Department of Gastrointestinal Surgery of the Qijiang People's Hospital, and to discuss the predictive effects of abdominal fat and muscle area on the short-term and long-term outcomes of gastric cancer patients after surgery.

1. Case collection Patients diagnosed with gastric cancer and undergoing radical gastric cancer surgery were screened according to the inclusion criteria. All patients had signed informed consent.

Inclusion criteria:

1. Diagnosed with gastric cancer by pathology or cytology;
2. Age >18 years;
3. Not having received chemotherapy, radiotherapy, targeted therapy or immunotherapy;
4. Patients with postoperative pathological stages other than stage IV, or without metastases in liver, lung or other distant organs confirmed by CT, MRI or B-ultrasound imaging and without surgical treatment;
5. Pre-operative CT examination data were kept in our hospital.

2. Data collection Collect patients' preoperative baseline information such as gender, age, body mass index (BMI), complications, tumor stage, etc. Collect patients' preoperative CT scans (make sure to include images from lumbar 1 to lumbar 5). Collect patients' surgical conditions such as operation time and intraoperative bleeding. Collect patients' postoperative complications during hospitalization; 3. Prognostic follow-up Closely follow up the death or cancer recurrence of patients after surgery. 4. Outcome indicators

1. Primary outcome indicators: overall survival (OS), disease-free survival (DFS), postoperative complications.
2. Secondary outcome indicators: postoperative recovery time, hospitalization time, postoperative weight change.

5. Image processing 3D Slicer was used to outline the range of subcutaneous fat, visceral fat, and muscle at the level of waist 1 to waist 5 on enhanced CT (5.0mm) images. Export the segmentation result as gpj.format, and select the Area Reading Calculator to calculate the area of fat and muscle at each level. Calculate fat area and muscle area at each level, calculate overall abdominal fat area and muscle area, and use the ratio of fat area to muscle area (e.g., visceral fat/skeletal muscle) as a predictor to generate the desired quantitative analyses.

6. Statistical Analysis

1. Basic characteristics and imaging indices were described as mean and standard deviation or median and standard deviation.
2. Univariate analysis including Kaplan-Meier survival analysis and Log-rank test were used to evaluate the effects of fat and muscle area on postoperative survival and complications.
3. Multivariate analysis including Cox regression models or Logistic regression models were used to evaluate the independent predictive role of abdominal fat and muscle area on surgical outcomes, controlling for potential confounders (e.g., age, gender, BMI, tumor stage, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of gastric cancer or colorectal cancer confirmed by pathology or cytology;
2. aged >18 years;
3. not received chemotherapy, radiotherapy, targeted therapy or immunotherapy;
4. post-operative pathological stages other than stage IV, or no liver, lung or other organs as confirmed by CT, MRI, B-ultrasound imaging.
5. patients who have pre-operative CT examination data kept in our hospital.

Exclusion Criteria:

1. Poor quality of preoperative CT images;
2. refusal to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients diagnosed with gastric and colorectal cancer and undergoing radical surgery for gastric and colorectal cancer at the study centre.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause or or loss to follow-up, whichever came first, assessed up to 60 months
  Overall survival was defined as time from date of diagnosis until the date of death from any cause or or loss to follow-up.

SECONDARY OUTCOMES:
Rate of postoperative complications | From date of surgery until the date of first documented postoperative complication, assessed up to 2 months after surgery.
  Surgical complications was defined as any postoperative complication occurring during the postoperative hospitalisation period.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - the First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - the Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Affiliated Yongchuan Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han J, Liu X, Tang M, Yang F, Ding Z, Wu G. Abdominal fat and muscle distributions in different stages of colorectal cancer. BMC Cancer. 2023 Mar 28;23(1):279. doi: 10.1186/s12885-023-10736-2. PMID 36978044
- [Background] Sun J, Lv H, Zhang M, Li M, Zhao L, Zeng N, Liu Y, Wei X, Chen Q, Ren P, Liu Y, Zhang P, Yang Z, Zhang Z, Wang Z. The Appropriateness Criteria of Abdominal Fat Measurement at the Level of the L1-L2 Intervertebral Disc in Patients With Obesity. Front Endocrinol (Lausanne). 2021 Dec 14;12:784056. doi: 10.3389/fendo.2021.784056. eCollection 2021. PMID 34970225
- [Background] Koh H, Hayashi T, Sato KK, Harita N, Maeda I, Nishizawa Y, Endo G, Fujimoto WY, Boyko EJ, Hikita Y. Visceral adiposity, not abdominal subcutaneous fat area, is associated with high blood pressure in Japanese men: the Ohtori study. Hypertens Res. 2011 May;34(5):565-72. doi: 10.1038/hr.2010.271. Epub 2011 Jan 13. PMID 21228782